CLINICAL TRIAL: NCT00143871
Title: Rituximab Plus High-dose Chemotherapy With Autologous Stem Cell Support for Non-Hodgkin's Lymphoma
Brief Title: Study of Rituximab Plus High-Dose Chemotherapy Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 0074
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Lymphoma, Non-Hodgkin's
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This study is being conducted to determine the safety, side effects, and response to a combination of an established high-dose chemotherapy regimen, plus the addition of Rituximab (which is a form of immunotherapy).

DETAILED DESCRIPTION:
Combination chemotherapy is the standard treatment as initial therapy for advanced stage aggressive Non-Hodgkin's lymphoma (NHL). Standard chemotherapy cures less than 40% of patients. When patients relapse, they may be eligible to receive high-dose chemotherapy with autologous stem cell support. Multiple studies have shown the value of high-dose chemotherapy, with increased disease-free survival and overall survival, when compared with second-line conventional chemotherapy. Unfortunately high-dose chemotherapy is curative in less than half the patients who receive it, and other treatment strategies are needed to improve the cure rate.

Another treatment option called immunotherapy is being tested in lymphoma patients. Immunotherapy involves attempts to use the immune system or products of the immune system to fight lymphoma. For example, NHL cells have a protein called CD20 on their surface. Rituximab is an antibody directed against the CD20 protein, which may result in the death of the lymphoma cell. Patients in this study will receive Rituximab to see if it is a safe treatment option for NHL patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, aggressive and/ or intermediate grade and high-grade B cell NHL, CD20 positive.
* In relapse after primary conventional chemotherapy
* Tumor sensitive (at least a partial response) to induction chemotherapy and/ or radiation therapy after treatment for relapse
* Treatment of CNS or meningeal disease (cytology-negative CSF) if present
* Treatment of CNS or meningeal disease (cytology-negative CSF) if present.
* Cumulative total doxorubicin dosage <500 mg/m2
* Performance score: 0-2
* Prior malignancies eligible if treated for cure and without active disease
* Patients must not be pregnant or nursing.
* Prior Immunotherapy is allowed
* Signed Informed Consent
* Absolute neutrophil count > 1500/ µl, platelet count >100,000/ µl
* Bilirubin <1.5 x normal, SGOT <2.5 x normal
* Serum creatinine <1.5 mg/dl
* Ejection fraction > 45% or > 40% with normal wall motion
* HIV negative
* FEV1, DLCO > 50% predicted

Exclusion Criteria:

* Pregnant or nursing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 2001-04; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Assess safety and toxicity after rituximab and high-dose chemotherapy

SECONDARY OUTCOMES:
Assess CD20 depletion in leukapheresis products after rituximab and high-dose chemotherapy, and monitor CD20 recovery post-transplant
Assess the response rate after rituximab and high-dose chemotherapy with autologous peripheral blood progenitor cell (PBPC) support, for patients with relapsed CD20+ Non-Hodgkin's lymphoma (NHL)
Assess progression-free and overall survival after rituximab and high-dose chemotherapy with PBPC support

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J. Hutchinson, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States